CLINICAL TRIAL: NCT04967482
Title: Drug-eluting Bead Transarterial Chemoembolization Compared With Conventional Transarterial Chemoembolization as the Conversion Therapy for Unresectable Large Hepatocellular Carcinoma: a Multicenter, Prospective, Nonrandomized Study
Brief Title: DEB-TACE vs. cTACE as Conversion Therapy for Unresectable Large HCC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIIR-06
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma Non-resectable
Keywords: Hepatocellular carcinoma; Transarterial chemoembolization; Conversion therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB-TACE (Experimental): DEB-TACE will be performed for the patients who choose DEB-TACE as the primary treatment.
  Interventions: Procedure: Drug-eluting bead transarterial chemoembolization (DEB-TACE)
- cTACE (Active Comparator): cTACE will be performed for the patients who choose cTACE as the primary treatment.
  Interventions: Procedure: Conventional transarterial chemoembolization (cTACE)

INTERVENTIONS:
Procedure: Drug-eluting bead transarterial chemoembolization (DEB-TACE) — The patients will receive DEB-TACE if they choose DEB-TACE as the primary treatment. DC Bead loaded with epirubicin (1 vial of DC Bead loaded with 60 mg of epirubicin) is used for chemoembolization. During follow-up, TACE will be repeated on demand based on the evaluation of the follow-up laboratory and imaging examination, and the technique method of each TACE procedure (i.e. DEB-TACE) for the same patient should be consistent.
  Arms: DEB-TACE
Procedure: Conventional transarterial chemoembolization (cTACE) — The patients will receive cTACE if they choose cTACE as the primary treatment. An emulsion of epirubicin in lipiodol wiil be injected into the tumor feeding artery. Afterwards, microspheres or polyvinyl alcohol particles mixed with contrast agent will be administered intraarterially until arterial flow stasis was achieved. Generally, the dose of lipiodol and epirubicin should not exceed 30 mL and 60 mg for each procedure. During follow-up, TACE will be repeated on demand based on the evaluation of the follow-up laboratory and imaging examination, and the technique method of each TACE procedure (i.e. cTACE) for the same patient should be consistent.
  Arms: cTACE

SUMMARY:
This study is conducted to evaluate the efficacy of drug-eluting bead transarterial chemoembolization (DEB-TACE) compared with conventional transarterial chemoembolization (cTACE) as the conversion therapy for unresectable large hepatocellular carcinoma (HCC).

DETAILED DESCRIPTION:
This is a multicenter, prospective and nonrandomized study to evaluate the efficacy of DEB-TACE (with DC Bead) compared with cTACE as the conversion therapy for unresectable large HCC.

At least 216 patients (≥ 108 patients in each arm) with initially unresectable large HCC (> 7cm) will be enrolled in this study. The patients will receive either DEB-TACE or cTACE as the primary treatment according to their won will. TACE can be repeated on demand based on the evaluation of follow-up laboratory and imaging examination by the multidisciplinary team, and the technique method of each TACE procedure (i.e. DEB-TACE or cTACE) for the same patient should be consistent. During follow-up, the potential resectability of the tumor will be assessed by the multidisciplinary team (MDT). Once the tumors become resectable, curative surgical resection will be recommended for the patients.

The primary end point of this study is success rate of conversion to resection. The secondary endpoints are objective response rate (ORR) of TACE, progression-free survival (PFS), times of TACE procedure to achieve conversion, conversion time, success rate of surgical resection, tumor recurrence rate after resection, tumor-free survival (TFS) of patients who undergo surgical resection, adverse events (AEs) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

1. Hepatocellular carcinoma confirmed by histopathology and/or cytology, or diagnosed clinically.
2. The tumor lesion was only localized in one liver lobe.
3. Large HCC with single lesion > 7 cm, or multiple lesions.
4. unresectable HCC evaluated by the surgeon team.
5. The patient is suitable for TACE treatment, which is evaluated by MDT.
6. At least one measurable intrahepatic target lesion.
7. Patients without cirrhosis, or with cirrhosis but the liver function of Child-Pugh Class A.
8. ECOG score of performance status ≤ 1 point.
9. Adequate organ and bone marrow function; the blood biochemical examination: platelet count ≥75×109/L, absolute value of neutrophils >1.5×109/L, hemoglobin ≥85 g/L, total bilirubin ≤30 μmol/L, albumin ≥35 g/L, ASL and AST≤5×ULN, creatinine≤1.5×ULN, INR<1.5 or PT/APTT normal range.
10. Patients have the willingness to receive TACE as the conversion therapy for surgical resection.

Exclusion Criteria:

1. Accompanied with tumor thrombus involving the main portal vein, first-order branch or bilateral branches of portal vein.
2. Accompanied with hepatic vein and vena cava tumor thrombus.
3. The extent of the lesion exceeds one liver lobe or extrahepatic metastasis.
4. Decompensated liver function, including: ascites, bleeding from gastroesophageal varices, and hepatic encephalopathy.
5. Those with organs (heart and kidneys) dysfunction who cannot tolerate TACE treatment and surgical hepatectomy.
6. History of other malignancies.
7. Uncontrollable infection.
8. Patients with active hepatitis B must undergo antiviral therapy to control HBV-DNA <10^3 IU/mL.
9. HCV patients need to complete the anti-HCV therapy before they are enrolled.
10. History of HIV.
11. Allergic to the drugs involved in the research.
12. Patients with gastrointestinal bleeding within 30 days, or other bleeding> CTCAE grade 3.
13. History of organ or cells transplantation. Previous treatment with TACE, intra-arterial infusion chemotherapy, radiotherapy, or systemic therapy
14. Those with bleeding tendency.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2021-07-09 (Actual); Primary Completion 2024-07-08 (Estimated); Study Completion 2024-07-08 (Estimated)

PRIMARY OUTCOMES:
Success rate of conversion to resection | 2 years.
  The proportion of patients with initially unresectable large HCC who were evaluated by the surgical team as suitable for second-stage surgical resection after TACE treatment.

SECONDARY OUTCOMES:
Objective response rate (ORR) of TACE treatment | 2 years.
  The percentage of patients who had a best overall tumor response rating of complete response (CR) or partial response (PR) which is assessed by the investigators according to modified Response Evaluaion Criteria in Solid Tumors (mRECIST).
Progression-free survival (PFS) | 3 years.
  The time between the first TACE treatment and the first occurrence of disease progression (PD) or death from any cause, whichever occurs first. For the patients who receive surgical resection after TACE, PD is defined as tumor recurrence/metastasis after resection. For the patients who did not undergo surgical resection, PD is assessed by the investigators according to mRECIST.
Times of TACE procedure to achieve conversion | 2 years.
  The number of TACE procedures performed for the patients when thier tumors become resectable. Resectability of the tumor is assessed by MDT during follow-up.
Time for successful conversion | 2 years.
  The duration between the first TACE treatment and the resectability of the tumor. Resectability is assessed by MDT.
Disease-free survival (TFS) of the patients who undergo resection | 2 years.
  The time between surgical resection and the first tumor recurrence/metastasis or death from any cause, whichever occurs first..
Adverse Events (AEs) | 3 years.
  Number of patients with AE, treatment-related AE (TRAE), serious adverse event (SAE), assessed by NCI CTCAE v5.0.
Overall survival (OS) | 3 years.
  The time from first TACE until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China